CLINICAL TRIAL: NCT05270616
Title: Robotic Versus Video-assisted Lobectomy/Segmentectomy for Lung Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Robotic lung ZYP
Record Dates: First submitted 2022-02-27; First posted 2022-03-08 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-02

CONDITIONS: Lung Diseases; Surgery
Keywords: robotic surgery; VATS; uniport; multiport
MeSH Terms: conditions — Lung Diseases | interventions — Robotic Surgical Procedures

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- robotic surgery group (Experimental): minimally invasive lung surgery using the Davinci robotic system to assist.
  Interventions: Procedure: robotic surgery
- uniport surgery group (Active Comparator): VATS minimally invasive lung surgery under the uniportal status.
  Interventions: Procedure: uniport surgery
- multiple- port surgery group (Active Comparator): VATS minimally invasive lung surgery under the multiple- port status.
  Interventions: Procedure: multiple- port surgery

INTERVENTIONS:
Procedure: robotic surgery — minimally invasive surgery using the Davinci robotic system
  Arms: robotic surgery group
Procedure: uniport surgery — VATS minimally invasive surgery under the uniportal status
  Arms: uniport surgery group
Procedure: multiple- port surgery — VATS minimally invasive surgery under the multiple- port status
  Arms: multiple- port surgery group

SUMMARY:
To compare the safety/efficacy of the robotic-assisted lobectomy/segmentectomy (RAL/S) with the video-assisted lobectomy/segmentectomy (VAL/S) for lung resection.

Video-assisted lobectomy/segmentectomy (VAL/S) for lung resection is divided into uniport group and multiple- port group.

ELIGIBILITY:
Inclusion Criteria:

1. good cardio- pulmonary function to tolerate surgery;
2. minimaly invasive surgery for lobectomy or segmentectomy or sleeve lobectomy;

Exclusion Criteria:

1. cardio- pulmonary function is not good enough to tolerate surgery;
2. huge tumor or extensive adhesion in thoracic cavity.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
mortality | 30 days after surgery
  incidence rate
conversion rate to open surgery | during surgery
  incidence rate
postoperative complications | within 7 days after surgery
  incidence rate
operation time | within 180 minutes
  minutes
duration of hospitalization | within 7 days after surgery
  days
days to tube removal | within 7 days after surgery
  days
retrieved lymph node | within 1 days after surgery
  amount
retrieved lymph node station | within 1 days after surgery
  amount
short- term PFS | 3 years
  proportion
short- term overall survival | 3 years
  proportion

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Hospital of Shandong University, Jinan, Shandong, China